CLINICAL TRIAL: NCT05899478
Title: Prospective, Multi-center, Randomized Controlled Study to Evaluate the Effectiveness and Safety of Suture-mediated Closure System Following Endovascular Peripheral Arterial Procedures
Brief Title: Suture-mediated Closure System Following Endovascular Peripheral Arterial Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Hengruihongyuan Medical Technology Co. LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPD01
Record Dates: First submitted 2023-05-05; First posted 2023-06-12 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Percutaneous Intervention Via Femoral Artery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tyknot® Suture-Mediated Closure System (Experimental): Arterial closure device used is Tyknot® Suture-Mediated Closure System
  Interventions: Device: Tyknot® Suture-Mediated Closure System
- Perclose® ProGlide Suture-Mediated Closure System (Active Comparator): Arterial closure device used is Perclose® ProGlide Suture-Mediated Closure System
  Interventions: Device: Perclose® ProGlide Suture-Mediated Closure System

INTERVENTIONS:
Device: Tyknot® Suture-Mediated Closure System — Arterial closure to ensure hemostasis at femoral artery puncture points
  Arms: Tyknot® Suture-Mediated Closure System
Device: Perclose® ProGlide Suture-Mediated Closure System — Arterial closure to ensure hemostasis at femoral artery puncture points
  Arms: Perclose® ProGlide Suture-Mediated Closure System

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of the suture-mediated closure system produced by Suzhou Hengrui Hongyuan Medical Technology Co., Ltd. following endovascular peripheral arterial procedures.

DETAILED DESCRIPTION:
Prospective, multi-center, randomized Comparative study using the Suture-mediated Closure System produced by Suzhou Hengrui Hongyuan Medical Technology Co., Ltd.as an investigational device and the Perclose® ProGlide Suture-Mediated Closure System as a comparator.

After going through the confirmation of inclusion/exclusion criteria with signed subjects, they will have a procedure either of the two devices. The subjects should follow designated physician's instructions accurately during the clinical trial period. There are about 4 times evaluations Including screening.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80
2. Patients who can use 5Fr to 21Fr sheath for common femoral artery puncture for interventional catheterization or therapy
3. Informed consent signed by the patient or legal representative

Exclusion Criteria:

1. Pregnancy or lactation period;
2. Diameter of femoral artery site for puncture< 5mm;
3. Have participated in another clinical study during the same period;
4. Known allergy to any device component, and/or contraindications of contrast agents and anticoagulants;
5. Vascular injury at the site of the approach;
6. Groin infection;
7. Morbid obesity (BMI≥40kg / ㎡);
8. Ultrasonographic assessment of the entire common femoral artery wall showed that the common femoral artery stenosis was ≥ 50%;
9. There are femoral aneurysms, arteriovenous fistulas or pseudoaneurysms in the common femoral artery;
10. Clamp vessel closures were used at the previous ipsilateral artery approach;
11. Hematoma at ipsilateral artery approach;
12. Other conditions deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Rate of successful hemostasis | 10 minutes
  Calculation method: Patients with successful hemostasis / total cases of subjects in the same group x 100%.
  Definition of successful hemostasis: Within 10 minutes after completion of the suturing procedure, there is no bleeding or hematoma at the puncture site, and no other intervention or surgical treatment is required.

SECONDARY OUTCOMES:
Operation time | Approximately 15-minutes after device removal
  The time for suturing with the vascular closure device. Definition of Operation time: The time it takes for the device to enter the artery, tie the knot, and then be successfully withdrawn from the vessel.
Hemostasis time | Approximately 15-minutes after compression
  The time from the catheter sheath is removed to compression is released and no bleeding occurs at the puncture site
Technical success rate | Approximately 15-minutes after device removal
  Calculation method: Patients with technical success/ total cases of subjects in the same group x 100%.
  Definition of Technical success: Successful placement of the device,smooth withdrawal, and completion fo the knot.
Evaluation of Compatibility with guidewires of the device | Approximately 15-minutes after device removal
  Scale from 1 point (worst) to 5 points (best)
Evaluation of Pushing performance of the device | Approximately 15-minutes after device removal
  Scale from 1 point (worst) to 5 points (best)
Evaluation of Withdrawal performance of the device | Approximately 15-minutes after device removal
  Scale from 1 point (worst) to 5 points (best)
Evaluation of Performance of tightening knot of the device | Approximately 15-minutes after device removal
  Scale from 1 point (worst) to 5 points (best)

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The First Affiliated Hospital of USTC, Hefei, Anhui
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Affiliated Hangzhou First People's Hospital ,Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Fourth Affiliated Hospital ,Zhejiang University School of Medicine, Yiwu, Zhejiang

IPD SHARING:
Plan to Share IPD: No